CLINICAL TRIAL: NCT04491669
Title: Screening of Gastrointestinal Tract Bleeding Causes Among Chronic Renal Failure Patients in Assuit University in a Single Study Center
Brief Title: Screening of Gastrointestinal Tract Bleeding Causes Among Chronic Renal Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Elsayed Mustafa Hussein Mandour, Dr., Assiut University
Other Study IDs: GIT bleeding among CKD
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: CKD; GIT - Gastrointestinal Tract Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Glomerular Filtration Rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: GFR - Glomerular Filtration Rate — Chronic Renal Failure staging according to GFR by Chronic Renal Failure EPI is:
  * Stage1 in which GFR>90 mil/min but evidence of kidney damage.
  * Stage 2 GFR 60-89 mil/min.
  * Stage 3 GFR 30-95 mil/min.
  * Stage 4 GFR 15-29 mil/min.
  * Stage 5 GFR<15 mil/min.

SUMMARY:
The aim of the current study is to screen different causes and characteristics of Gastrointestinal bleeding in Chronic Renal Failure patients at Assuit University Hospital according to their stages based on e GFR (Stage I to IV), in order to assess different modalities of therapeutic intervention from medical therapy up to therapeutic intervention.

DETAILED DESCRIPTION:
* Chronic Renal Failure is defined as presence of reduced glomerular filtration rate (GFR) < 60 ml/min/ 1.73 m2 and/or evidence of kidney damage (usually indicated by albuminuria or proteinuria) for > 3 months or more irrespective of cause (Kiapidou et al., 2019).
* Chronic Renal Failure stages are classified according to the National Kidney Foundation in to five stages according to estimated GFR (Ikizler 2009).
* The prevalence of Chronic Renal Failure is continuously rising in concert with the rising epidemic of its risk factors including ageing, diabetes, obesity, metabolic syndrome, smoking, and hypertension (Stevens and Levin 2013).
* Gastrointestinal bleeding, is all forms of bleeding in the gastrointestinal tract, from the mouth to the rectum. When there is significant blood loss over a short time, symptoms may include vomiting red blood, vomiting black blood, bloody stool, or black stool. Small amounts of bleeding over a long time may cause iron-deficiency anemia resulting in feeling tired or heart-related chest pain.

Other symptoms may include abdominal pain, shortness of breath, pale skin, or passing out. Sometimes in those with small amounts of bleeding no symptoms may be present. (Bong Sik Matthew Kim. 2014)

• Preliminary data suggest an association between Chronic Renal Failure and Gastrointestinal Bleeding. Individuals with even mild to moderate Chronic Renal Failure warrant clinical attention regarding the risk of hospitalization with Gastrointestinal bleeding. (Kunihiro Matsushita, 2016 Oct 7) reported that the prevalence of Gastrointestinal bleeding was significantly higher in patients with Chronic Renal Failure compared to patients without Chronic Renal Failure.

ELIGIBILITY:
Inclusion Criteria:

* One hundred Chronic Renal Failure patients with different stages (stage I to IV) according to the National Kidney Foundation are recruited from inpatients of renal unit in internal medicine department, Assuit university hospitals. Their GFR will assessed by using Chronic Renal Failure EPI equation measured as GFR=166 x(s cr/0.7)-1.209X(0.993)age if female, and GFR=163X(s cr/0.9)-1.209x(0.993)age if male. (Andrews et al 2008).

Chronic Renal Failure staging according to GFR by Chronic Renal Failure EPI is:

* Stage1 in which GFR>90 mil/min but evidence of kidney damage.
* Stage 2 GFR 60-89 mil/min.
* Stage 3 GFR 30-95 mil/min.
* Stage 4 GFR 15-29 mil/min.
* Stage 5 GFR<15 mil/min.

Exclusion Criteria:

* All Patients with local causes of Gastrointestinal Bleeding

  * Benign and Malignant tumors in Gastrointestinal Tract.
  * Patients with Hemorrhoids or anal fissures.
  * Patients with Mallory-Weiss tears.
  * patients with Diverticular disease.
  * patients with Colon polyps.
  * patients with infectious causes of GIT bleeding (Salmonella, Shigella)
  * patients with Angiodysplasia.
  * patients with Esophageal varices

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic Renal Failure patients with different stages (stage I to IV) according to the National Kidney Foundation are recruited from inpatients of renal unit in internal medicine department, Assuit university hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of different modalities of therapeutic intervention. | one year from October 2020 to October 2021
  medical therapy up to therapeutic intervention data will be received.

CONTACTS AND LOCATIONS:
Overall Officials: Effat AH Tony, Prof. Dr., Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barkun AN, Bardou M, Kuipers EJ, Sung J, Hunt RH, Martel M, Sinclair P; International Consensus Upper Gastrointestinal Bleeding Conference Group. International consensus recommendations on the management of patients with nonvariceal upper gastrointestinal bleeding. Ann Intern Med. 2010 Jan 19;152(2):101-13. doi: 10.7326/0003-4819-152-2-201001190-00009. PMID 20083829
- [Background] Zuccaro G Jr. Management of the adult patient with acute lower gastrointestinal bleeding. American College of Gastroenterology. Practice Parameters Committee. Am J Gastroenterol. 1998 Aug;93(8):1202-8. doi: 10.1111/j.1572-0241.1998.00395.x. No abstract available. PMID 9707037
- [Background] Kim BS, Li BT, Engel A, Samra JS, Clarke S, Norton ID, Li AE. Diagnosis of gastrointestinal bleeding: A practical guide for clinicians. World J Gastrointest Pathophysiol. 2014 Nov 15;5(4):467-78. doi: 10.4291/wjgp.v5.i4.467. PMID 25400991
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Ishigami J, Matsushita K. Clinical epidemiology of infectious disease among patients with chronic kidney disease. Clin Exp Nephrol. 2019 Apr;23(4):437-447. doi: 10.1007/s10157-018-1641-8. Epub 2018 Sep 3. PMID 30178234